CLINICAL TRIAL: NCT06458348
Title: Construction and Empirical Study of Local Opera Appreciation Combined With Medical Gymnastics Training Program for Elderly Patients With Post-stroke Cognitive Impairment
Brief Title: Local Opera Viewing Combined Medical Gymnastics for Elderly PSCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhangzhou Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Zhangzhou Municipal Hospital
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Post-stroke Cognitive Impairment

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Local opera appreciating (Experimental): Received the local drama viewing .When the PSCI patient was hospitalized and discharged for 12 weeks. appreciating local drama for 30-45 minutes every day
  Interventions: Behavioral: Local opera appreciating and Medical gymnastics training
- Medical gymnastics training (Experimental): Conducted medical gymnastics training .When the PSCI patient was hospitalized and discharged for 12 weeks. conduct medical gymnastics training for 30-45 minutes every day
  Interventions: Behavioral: Local opera appreciating and Medical gymnastics training
- Local opera appreciating and Medical gymnastics training (Experimental): Received the drama viewing and conducted the medical gymnastics training .When the PSCI patient was hospitalized and discharged for 12 weeks. Appreciating local drama for 30-45 minutes and conduct medical gymnastics training for 30-45 minutes every day
  Interventions: Behavioral: Local opera appreciating and Medical gymnastics training
- Routine treatment (No Intervention): When the PSCI patient was hospitalized and discharged for 12 weeks, Received the routine treatment and care.

INTERVENTIONS:
Behavioral: Local opera appreciating and Medical gymnastics training — To construct a local opera viewing combined medical gymnastics training program for elderly patients with post-stroke cognitive impairment, and to explore its feasibility, acceptability and safety.
  Arms: Local opera appreciating; Local opera appreciating and Medical gymnastics training; Medical gymnastics training

SUMMARY:
local opera viewing combined medical gymnastics for elderly PSCI

DETAILED DESCRIPTION:
Cognitive impairment and hemiplegia are the two major problems faced by elderly patients with cognitive impairment after stroke. The application of local drama viewing and combined medical gymnastics training aims to improve sports and cognitive function. Local drama viewing and medical gymnastics training integrates drama art cognition and medical sports, is a beneficial scientific attempt.

To construct a local opera viewing combined medical gymnastics training program for elderly patients with post-stroke cognitive impairment, and to explore its feasibility, acceptability and safety.

ELIGIBILITY:
Inclusion Criteria:

Stroke patients who were hospitalized in the Department of Neurology of Zhangzhou Hospital and met the PSCI diagnostic criteria of the Expert Consensus on the Prevention and Treatment of Cognitive Impairment after Stroke in China were the subjects of the study. ① Stroke patients confirmed by neuroimaging, onset time within 1 week; (2) Cognitive impairment occurs after stroke events; ③ The scores of the simple mental state examination scale were points in the illiterate group, points in the primary school group, points in the secondary school group, and points in the college group; ④ can maintain independent sitting position ≥30 min; ⑤ Age ≥60 years old; ⑥ Volunteer to join the study and receive intervention treatment.

Exclusion Criteria:

* Other causes affect or lead to cognitive impairment, such as consciousness disorder, malignant tumor, severe liver and kidney insufficiency; ② There are serious cardiopulmonary and other systemic diseases; Visual or hearing impairment; ④ have emotional behavior abnormalities and mental illness (including depression); ⑤ A history of alcohol or drug abuse

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
NIH stroke scale, NIHSS | Before and at 3 months after the intervention
  NIHSS is based on structural neurological examination and gives a score between 0 and 42. Higher scores indicate a more severe neurological deficit . The NIHSS-score 5 indicates mild neurological deficit, and 5 to 15 indicates moderate neurological deficit score> 20 generally considered to indicate "severe" stroke, whereas patients with isolated severe aphasia (NIHSS score 2 or 3) may have damaging . Nerve deficit (NIHSS) , which involves 15 factors such as movement, sensory, visual field, and the score range from 0 to 42. The deficit is divided into three grades: mild, moderate and severe, respectively 0-15,16~30 and 31~42 points.
Muscle strength | Before and at 3 months after the intervention
  When level 6 (level 0~5) muscle strength recording method, let the patient do the muscle contraction movement in turn, the examiner give resistance, or When the patient was instructed to maintain a position, the examiner tried to change the position to determine muscle strength (Table 4-3). Six-level recording method of attack 4-3 muscle strength
  Level 0 Complete paralysis, with no muscle contraction Level 1 Muscles can contract, but can not act Level 2 The limb can move on the bed surface, but can not resist their own gravity, that is, can not lift Level 3 The limb can resist gravity off the bed surface, but can not resist resistance Level 4 The body can do antiresistance movements, but not completely Level 5 Normal muscle strength
Montreal cognitive assessment, MoCA-Beijing | Before and at 3 months after the intervention
  The version includes eight aspects of cognitive domain test: memory, visual space, execution, attention, computing, language, time orientation, location orientation, total score of 30 points, the higher the score, the cognitive function of the better, the illiterate group 13 points, elementary school group 19 points, junior high school and above test 24 points can be judged as impaired cognitive function impaired , to correct the cultural bias. MoCA, specifically designed for screening MCI, has high sensitivity (80% to 100%) and specificity (50% to 7 6%) in identifying MCI.
Mini-Mental State Examination, MMSE | Before and at 3 months after the intervention
  MMSE is the first simple tool compiled by Folstein et al. to assess cognitive function. After practice, it is gradually used for screening of dementia patients, judge the severity of cognitive impairment and track the changes of the condition. Its sensitivity in dementia screening diagnosis is 80-90% and specificity is 70-80% . The scale covers cognitive domains such as directional force, memory, attention and calculation, speech, and visual space. The scale has 30 entries with a total score of 30, which can be graded according to MMSE, with 21 to 26 mild dementia, 11 to 20 moderate dementia, and 0 to 10 severe dementia . This study adopted the version revised by domestic scholar Wang Zhengyu et al. , with 30 items and a total of 30 points. The abnormal score was divided into 17 points for illiterate group, 20 points in primary school group and 24 points in middle school and above group. AD patients with this scale was excluded in this study.

SECONDARY OUTCOMES:
Hamilton Anxiety Rating Scale | Before and at 3 months after the intervention
  The Hamilton Anxiety Scale (Hamilton Anxiety Scale, HAMA) is the most clinically used to assess anxiety symptoms in adults For a wide range of his evaluation tools.14 items, using 5 grades ranging from 0 to 4. Higher scores indicate greater anxiety.
Hamilton Depression Rating Scale | Before and at 3 months after the intervention
  The Hamilton Depression Scale (Hamilton DepressionScaleHAMD) clinically evaluates depressive symptoms in adults .The most widely used evaluation tools. There are three versions of 17 items, 21 items, and 24 items. Most of the items use 5 grades of 0 to 4, but a few Grade 3 score from 0 to 2. Higher scores indicate greater depression.
Pittsburgh Sleep Quality Index | Before and at 3 months after the intervention
  MMSE is the first simple tool compiled by Folstein et al. to assess cognitive function. After practice, it is gradually used for screening of dementia patients, judge the severity of cognitive impairment and track the changes of the condition. Its sensitivity in dementia screening diagnosis is 80-90% and specificity is 70-80% . The scale covers cognitive domains such as directional force, memory, attention and calculation, speech, and visual space. The scale has 30 entries with a total score of 30, which can be graded according to MMSE, with 21 to 26 mild dementia, 11 to 20 moderate dementia, and 0 to 10 severe dementia [93]. This study adopted the version revised by domestic scholar Wang Zhengyu et al. [69], with 30 items and a total of 30 points. The abnormal score was divided into 17 points for illiterate group, 20 points in primary school group and 24 points in middle school and above group. AD patients with this scale was excluded in this study.
Stroke Impact Scale，SIS | Before and at 3 months after the intervention
  In order to evaluate how much stroke affects PSCI health and life, to know the PSCI own views on the impact of stroke. questions about the dysfunction caused by stroke and the impact on the life of PSCI
Subscales of the Functional Assessment of Communication Skills, SFACS | Before and at 3 months after the intervention
  SFACS was developed by Frattali et al in 1995 .2015 Chinese by Chen Huiying. This scale was originally used in patients with aphasia, and was later widely used by other scholars in dementia, stroke, brain trauma and other fields. It evaluates the communication functions from four domains , Each domain has four qualitative dimensions. There are 43 entries in this scale, which takes about 20 minutes, and the scoring standard is a 7-point system: 1= not completed, 2= need a large amount of assistance, 3 = general to large amount of assistance, 4= general assistance, 5 = small amount to general assistance, 6= small amount of assistance, 7 = completed independently. FACS can evaluate communication skills using either the total questionnaire or subscales, with higher scores indicating better communication skills.

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Xiao, MSc, Principal Investigator — Zhangzhou Municipal Hospital